CLINICAL TRIAL: NCT05761613
Title: Ceragenin Coated Endotracheal Tubes for the Eradication of Ventilator Associated Pneumonia - A Prospective, Longitudinal, Cross-over, Interrupted Time, Implementation Study (CEASE VAP Study)
Brief Title: Ceragenin Coated Endotracheal Tubes for the Prevention of Ventilator Associated Pneumonia
Acronym: CEASEVAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. John Muscedere (Other)
Responsible Party: Sponsor-Investigator, Dr. John Muscedere, Professor of Medicine, Queen's University
Organization: Queen's University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 6036323
Record Dates: First submitted 2023-02-23; First posted 2023-03-09 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All pneumonia outcomes will be adjudicated by a panel blinded to allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Endotracheal Tube with Subglottic Secretion Drainage (Active Comparator): All patients in this arm will be intubated with an ETT with subglottic secretion drainage
  Interventions: Device: Endotracheal tube with subglottic secretion drainage
- CeraShield Endotracheal Tube (Active Comparator): All patients in this arm will be intubated with a ceragenin coated ETT
  Interventions: Device: CeraShield Endotracheal Tube

INTERVENTIONS:
Device: CeraShield Endotracheal Tube — An endotracheal tube coated with with an antimicrobial hydrophilic coating containing ceragenins (CSAs)
  Arms: CeraShield Endotracheal Tube
Device: Endotracheal tube with subglottic secretion drainage — An endotracheal tube with subglottic secretion drainage
  Arms: Endotracheal Tube with Subglottic Secretion Drainage

SUMMARY:
Critically ill patients are at high risk of acquiring pneumonia during the time that they are mechanically ventilated. This is known as ventilator-associated pneumonia (VAP). VAP results in increased duration of mechanical ventilation, increased ICU and hospital stay, increased risk of death and increased health care costs. VAP occurs in 20% of patients and it is estimated that each case of VAP costs the health care system $10 to 15,000 Canadian. Because of its impact on patient outcomes and the health care system, VAP is regarded as an important patient safety issue and there is an urgent need for better prevention strategies.

Invasive mechanical ventilation requires the passage of an endotracheal tube (ETT) through the pharynx which is frequently colonized with bacterial pathogens and a bio-film rapidly forms on the ETT. VAP results either from aspiration of contaminated oropharyngeal secretions or from aspiration of bacteria from the bio-film. In this project, the efficacy of a novel ETT coated with an antibiotic compound that has been shown to reduce the formation of bio-film and pathogen colonization will be tested. Preliminary evidence as to whether utilization of this novel ETT reduces the occurrence of VAP and improves patient outcomes will be obtained through the conduct of a pragmatic, prospective, longitudinal, interrupted time, cross-over implementation study.

DETAILED DESCRIPTION:
The innovation that is being studied is a novel antibiotic coated endotracheal tube (ETT) for the prevention of ventilator associated pneumonia (VAP) in critically ill, mechanically ventilated patients. The novel ETT is the CeraShield ETT consisting of a standard ETT with an antimicrobial hydrophilic coating containing ceragenins (CSAs) on the inner and outer lumen of the device, as well as the inflatable cuff. The CSA coating on the CeraShield protects it from microbial colonization and bio-film growth. The CSA ETT is otherwise equivalent to standard ETT tubes currently in use and is licensed in Canada for clinical use as a Class 2 device.

1. It is hypothesized that CSA coated ETTs will reduce the incidence of Ventilator Associated Pneumonia and improve clinical outcomes including antibiotic utilization when compared to ETTs currently in use.
2. It is hypothesized that a definitive cluster randomized multi-center study is feasible and supported by the data from this study.

To test the hypotheses, an Interrupted Time Series Cross-Over Implementation Study will be used to provide preliminary evidence of the efficacy of the CeraShield ETT compared to the ETT currently used at the study center in critically ill mechanically ventilated patients. This study will inform and be modified to conduct a future large multi-center cluster randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Adult critically ill patients with respiratory failure requiring intubation

Exclusion Criteria:

1. Admission to hospital or ICU with a non-study ETT already in place
2. Presence of a tracheostomy on ICU admission
3. Unable to be intubated with non-study ETT
4. Declined participation in research or data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Ventilator Associated Pneumonia | Admission to within 48 hours of cessation of invasive mechanical ventilation or 28 days
  The primary outcome will be the occurrence of VAP defined as new, progressive, or persistent radiographic infiltrate on chest radiograph plus any 2 of the following: (1) fever (core temperature >38°C) or hypothermia (temperature <36°C); (2) white blood cell count less than 3.0 × 106/L or exceeding 10 × 106/L, and (3) purulent sputum

SECONDARY OUTCOMES:
Antibiotic Utilization | 28 days after intubation
  Antibiotic free days defined as alive and not recieving antibiotics in the 28 day period after intubation
Health care utilization | 90 days
  Duration of mechanical ventilation, duration of ICU stay, duration of hospital stay
Health care utilization | 28 days
  Ventilator Free Days defined as alive and off ventilation in the 28 day period after intubation
Hospital Mortality | 90 days
  Mortality while hospitalized
Airway outcomes | Within 48 hours of extubation
  Incidence of post-extubation stridor, lack of endotracheal tube cuff leak
Re-intubation | Within 48 hours of extubation
  Rate of re-intubation after extubation from invasive mechanical ventilation
Acceptability of the Intervention | During the conduct of the trial up to 1 year from study initiation
  Measured by the Acceptability of Intervention Measure Tool (AIM). AIM is a 5 point scale that measures the perception of implementation stakeholders that a new treatment (in this study new type of ETT) is agreeable or satisfactory. AIM is an ordinal scale that ranges from completely agree to completely disagree.
Feasibility of multi-center cluster randomized trial - 1 | During the trial up to 1 year from study start
  Determination of required sample size for a multi-center study based on the event rates (Occurrence of VAP as in outcome 1 and antibiotic utilization as in outcome 2) in this single center trial. Sample size will be calculated for the multicenter study and feasibility will be informed by the magnitude of the sample size and the potential resources required to conduct such as study including the number of centers.
Feasibility of multi-center cluster randomized trial - 2 | During the trial up to 1 year from study start
  Acceptable availability of routinely collected data for analysis of study conduct defined as less than 10% missing data

CONTACTS AND LOCATIONS:
Overall Officials: John MUSCEDERE, MD, Principal Investigator — Queens University
Locations (1):
- Kingston Health Sciences Center, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Safdar N, Dezfulian C, Collard HR, Saint S. Clinical and economic consequences of ventilator-associated pneumonia: a systematic review. Crit Care Med. 2005 Oct;33(10):2184-93. doi: 10.1097/01.ccm.0000181731.53912.d9. PMID 16215368
- [Background] Muscedere JG, Day A, Heyland DK. Mortality, attributable mortality, and clinical events as end points for clinical trials of ventilator-associated pneumonia and hospital-acquired pneumonia. Clin Infect Dis. 2010 Aug 1;51 Suppl 1:S120-5. doi: 10.1086/653060. PMID 20597661
- [Background] Muscedere J, Rewa O, McKechnie K, Jiang X, Laporta D, Heyland DK. Subglottic secretion drainage for the prevention of ventilator-associated pneumonia: a systematic review and meta-analysis. Crit Care Med. 2011 Aug;39(8):1985-91. doi: 10.1097/CCM.0b013e318218a4d9. PMID 21478738
- [Background] Diaconu O, Siriopol I, Polosanu LI, Grigoras I. Endotracheal Tube Biofilm and its Impact on the Pathogenesis of Ventilator-Associated Pneumonia. J Crit Care Med (Targu Mures). 2018 Apr 1;4(2):50-55. doi: 10.2478/jccm-2018-0011. eCollection 2018 Apr. PMID 30581995
- [Background] Epand RM, Epand RF, Savage PB. Ceragenins (cationic steroid compounds), a novel class of antimicrobial agents. Drug News Perspect. 2008 Jul-Aug;21(6):307-11. doi: 10.1358/dnp.2008.21.6.1246829. PMID 18836587
- [Background] Grimshaw J, Campbell M, Eccles M, Steen N. Experimental and quasi-experimental designs for evaluating guideline implementation strategies. Fam Pract. 2000 Feb;17 Suppl 1:S11-6. doi: 10.1093/fampra/17.suppl_1.s11. PMID 10735262
- [Derived] Symonds NE, Meng EXM, Boyd JG, Boyd T, Day A, Hobbs H, Maslove DM, Norman PA, Semrau JS, Sibley S, Muscedere J. Ceragenin-coated endotracheal tubes for the reduction of ventilator-associated pneumonia: a prospective, longitudinal, cross-over, interrupted time, implementation study protocol (CEASE VAP study). BMJ Open. 2024 Feb 2;14(2):e076720. doi: 10.1136/bmjopen-2023-076720. PMID 38309761